CLINICAL TRIAL: NCT02470013
Title: Medical and Health Economic Benefit of Oral Nutritional Supplements (ONS) in Ambulant Patients
Acronym: ECONONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfrimmer Nutricia GmbH, Erlangen , Germany (Industry)
Responsible Party: Principal Investigator, Kristina Norman, PD Dr. Kristina Norman, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECONONS
Record Dates: First submitted 2015-01-14; First posted 2015-06-12 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Malnutrition
Keywords: Malnutrition; Geriatrics; Enteral Nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Nutrition counselling and balanced, energy dense, moderate protein sip feed ('Fortimel Compact, Nutricia GmbH) for 3 months
  Interventions: Dietary Supplement: Balanced, energy dense, moderate protein sip feed
- Control Group (No Intervention): Nutrition counselling upon hospital discharge (usual care)

INTERVENTIONS:
Dietary Supplement: Balanced, energy dense, moderate protein sip feed — 2x 125 ml bottles (equiv. 600 kcal) of Fortimel Compact daily for 3 months in addition to normal eating habits
  Arms: Intervention Group

SUMMARY:
The aim of this study is to assess the benefit of a 3-month intervention with oral nutritional supplements (ONS) in older ambulant patients with reference to functional limitations and quality of life as well as the consumption of health care resources.

DETAILED DESCRIPTION:
Study participants are assessed upon discharge from the hospital and again after 3 months. Upon discharge all patients receive nutrition counselling with special focus on an energy rich diet. Additionally, the intervention group receives ONS. The investigators hypothesize an improvement in functional limitations and health economic benefits due to the post-hospital nutritional intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Informed written consent
* Independent community dwelling after discharge
* Existing or risk of malnutrition
* Normal cognitive status according to Mini-Mental State Examination (MMSE ≥ 24 points)
* Life expectancy of > 3 months according to treating doctor
* No severe heart disease (New York Heart Association (NYHA) functional classification of 3+), liver disease (Child Pugh Score = A, B) or kidney insufficiency (glomerular filtration rate < 30 ml/min)
* No chemo or radiation therapy
* No derailed diabetes mellitus or metabolic decompensation

Exclusion Criteria:

* Age < 60 years
* Lack of informed written consent
* Dependent living conditions after discharge
* No risk of malnutrition
* Low cognitive status according to Mini-Mental State Examination (MMSE < 24 points)
* Life expectancy of < 3 months according to treating doctor
* Severe heart disease (New York Heart Association (NYHA) functional classification of 3+), liver disease (Child Pugh Score = C) or kidney insufficiency (glomerular filtration rate < 30 ml/min)
* Chemo or radiation therapy
* Derailed diabetes mellitus or metabolic decompensation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-11; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in functional limitations and activities of daily living (single validated questionnaire) | Baseline (hospital discharge) and after 3 months

SECONDARY OUTCOMES:
Functional Parameter: timed up & go | Baseline (hospital discharge) and after 3 months
Functional Parameter: stair climbing | Baseline (hospital discharge) and after 3 months
Functional Parameter: lung function | Baseline (hospital discharge) and after 3 months
Functional Parameter: gait analysis | Baseline (hospital discharge) and after 3 months
Strength Parameter: Hand grip strength | Baseline (hospital discharge) and after 3 months
Strength Parameter: Knee extension strength | Baseline (hospital discharge) and after 3 months
Quality of life (validated questionnaire) | Baseline (hospital discharge) and after 3 months
Body composition (bioelectric impedance analysis) | Baseline (hospital discharge) and after 3 months
Consumption of health care resources (questionnaire) and cost analysis | From baseline (hospital discharge) during subsequent 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Norman, PD Dr., Principal Investigator — Charite Research Group on Geriatrics
Locations (1):
- Charite University Medicine, Research Group on Geriatrics, Berlin, Germany

REFERENCES:
- [Background] Norman K, Pirlich M, Smoliner C, Kilbert A, Schulzke JD, Ockenga J, Lochs H, Reinhold T. Cost-effectiveness of a 3-month intervention with oral nutritional supplements in disease-related malnutrition: a randomised controlled pilot study. Eur J Clin Nutr. 2011 Jun;65(6):735-42. doi: 10.1038/ejcn.2011.31. Epub 2011 Mar 16. PMID 21407248
- [Background] Norman K, Kirchner H, Freudenreich M, Ockenga J, Lochs H, Pirlich M. Three month intervention with protein and energy rich supplements improve muscle function and quality of life in malnourished patients with non-neoplastic gastrointestinal disease--a randomized controlled trial. Clin Nutr. 2008 Feb;27(1):48-56. doi: 10.1016/j.clnu.2007.08.011. Epub 2007 Oct 25. PMID 17964008
- [Background] Neelemaat F, Bosmans JE, Thijs A, Seidell JC, van Bokhorst-de van der Schueren MA. Oral nutritional support in malnourished elderly decreases functional limitations with no extra costs. Clin Nutr. 2012 Apr;31(2):183-90. doi: 10.1016/j.clnu.2011.10.009. Epub 2011 Nov 8. PMID 22071290